CLINICAL TRIAL: NCT02487966
Title: Optimizing Rehabilitation for Phantom Limb Pain Using Mirror Therapy and Transcranial Direct Current Stimulation (tDCS)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Spaulding Rehabilitation Hospital (Other)
Collaborators: Massachusetts Eye and Ear Infirmary (Other)
Responsible Party: Principal Investigator, Felipe Fregni, MD, PhD, MPH, Principal Investigator, Spaulding Rehabilitation Hospital
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: 2015P001065
Record Dates: First submitted 2015-06-22; First posted 2015-07-02 (Estimated); Results first posted 2021-06-21 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Phantom Limb Pain; Amputation, Traumatic
Keywords: tDCS; Mirror Therapy; Phantom Limb Pain; Traumatic amputation
MeSH Terms: conditions — Phantom Limb; Amputation, Traumatic | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (4):
- Active tDCS and Active Mirror Therapy (Experimental): Subjects will receive 20 minutes of active tDCS, while receiving 15 minutes of active Mirror Therapy.
  Interventions: Device: transcranial Direct Current Stimulation (tDCS): active (Soterix ©); Behavioral: Mirror Therapy: active
- Active tDCS and sham Mirror Therapy (Experimental): Subjects will receive 20 minutes of active tDCS, while receiving 15 minutes of sham Mirror Therapy.
  Interventions: Device: transcranial Direct Current Stimulation (tDCS): active (Soterix ©); Behavioral: Mirror Therapy: Sham
- Sham tDCS and active Mirror Therapy (Experimental): Subjects will receive 20 minutes of sham tDCS, while receiving 15 minutes of active Mirror Therapy.
  Interventions: Behavioral: Mirror Therapy: active; Device: transcranial Direct Current Stimulation (tDCS): sham (Soterix ©)
- Sham tDCS and sham Mirrory Therapy (Sham Comparator): Subjects will receive 20 minutes of sham tDCS, while receiving 15 minutes of sham Mirror Therapy.
  Interventions: Device: transcranial Direct Current Stimulation (tDCS): sham (Soterix ©); Behavioral: Mirror Therapy: Sham

INTERVENTIONS:
Device: transcranial Direct Current Stimulation (tDCS): active (Soterix ©) — Subjects will undergo tDCS stimulation. For both active and sham stimulation, we will use electrodes of 35cm^2, at an intensity of 2mA on the primary motor cortex contralateral to the amputated leg. For active tDCS, the subject will undergo stimulation for 20 minutes.
  Arms: Active tDCS and Active Mirror Therapy; Active tDCS and sham Mirror Therapy
Behavioral: Mirror Therapy: active — Subjects will be asked to perform movements (15 minutes daily) using the unaffected limb while watching its mirrored reflection superimposed over the affected limb. During Mirror Therapy, subjects will be asked to consciously relate the movement observed in the mirror to their phantom limb and to keep their attention focused on the task. Instructions will be explained verbally, demonstrated by a therapist, and performed by the subject in front of the therapist.
  Arms: Active tDCS and Active Mirror Therapy; Sham tDCS and active Mirror Therapy
Device: transcranial Direct Current Stimulation (tDCS): sham (Soterix ©) — Subjects will undergo tDCS stimulation. For both active and sham stimulation, we will use electrodes of 35cm^2, at an intensity of 2mA on the primary motor cortex contralateral to the amputated leg. The subject will undergo stimulation for 20 minutes. This is the same parameters as the active one, except the current will be ramped up and then down again (for 30 seconds total) to simulate the feeling of active stimulation.
  Arms: Sham tDCS and active Mirror Therapy; Sham tDCS and sham Mirrory Therapy
Behavioral: Mirror Therapy: Sham — Subjects will be asked to perform movements (15 minutes daily) using the unaffected limb while watching its mirrored reflection superimposed over the affected limb, only the mirror will be covered. During Mirror Therapy, subjects will be asked to consciously relate the movement observed in the mirror to their phantom limb and to keep their attention focused on the task. Instructions will be explained verbally, demonstrated by a therapist, and performed by the subject in front of the therapist. We will use the same all of these techniques as active Mirror Therapy only the mirror will be covered during all activities.
  Arms: Active tDCS and sham Mirror Therapy; Sham tDCS and sham Mirrory Therapy

SUMMARY:
This is a two-site study that explores the effects of mirror therapy and transcranial Direct Current Stimulation (tDCS, Soterix ©) in a randomized factorial controlled trial in which patients will be assigned to one of four groups: active tDCS and active MT; sham tDCS and active MT; active tDCS and sham MT (which consists of using a covered mirror for the therapy); and both sham tDCS and sham MT (covered mirror).

DETAILED DESCRIPTION:
Phantom limb pain (PLP) belongs to a group of neuropathic pain syndromes that is characterized by pain in the amputated limb. Rehabilitation for chronic pain involves a structured treatment plan targeting all dimensions of the pain experience, and should include a comprehensive interdisciplinary approach that allows patients to receive the most benefit according to their needs. As in other chronic pain syndromes, chronic Phantom limb pain (PLP) is often difficult to treat; showing to be resistant to classical pharmacological and surgical treatment approaches.

In this context, we hypothesize that novel treatments of PLP need to target specific neural networks associated with this maladaptive plasticity. Transcranial direct current stimulation (tDCS,Soterix ©) is a powerful and non-invasive technique of brain stimulation that is known to significantly modulate plasticity and alleviate chronic pain in various syndromes. device for this trial. This study usiGiven tDCS underlying neural mechanisms, it is critical to use a multimodal approach to treatment - using both tDCS and behavioral therapy simultaneously. In this case, an ideal therapy is mirror therapy (MT).

Recently, we showed that anodal tDCS can induce a selective short-lasting relief from PLP, and repeated applications of anodal tDCS induces long-lasting analgesic effects. These preliminary results show that tDCS may be a promising rehabilitative tool for the management of chronic PLP. This neurorehabilitation technique is commonly used in PLP, and is designed to modulate cortical mechanisms of pain by performing movements using the unaffected limb in front of a mirror. We propose to carry out a mechanistic, factorial, randomized controlled trial to evaluate a novel rehabilitation approach combining tDCS and MT in PLP patients. We aim to compare the brain changes before and after treatment in order to study the mechanisms underlying PLP.

ELIGIBILITY:
Inclusion Criteria:

1. Able to provide informed consent to participate in the study.
2. Subject is older than 18 years.
3. Unilateral lower limb amputation.
4. Traumatic amputation greater than 1 year ago.
5. Chronic PLP for at least 3 months previous to enrollment in the study, experienced regularly for at least once a week.
6. Average pain of at least 4 on a numeric rating scale in the previous week (NRS; ranging from 0 to 10).
7. If the subject is taking any medications, dosages must be stable for at least 2 weeks prior to the enrollment of the study.

Exclusion Criteria:

1. Pregnancy or trying to become pregnant in the next 2 months.
2. History of alcohol or drug abuse within the past 6 months as self-reported.
3. Presence of the following contraindication to transcranial direct current stimulation and transcranial magnetic stimulation

   * Ferromagnetic metal in the head (e.g., plates or pins, bullets, shrapnel)
   * Implanted neck or head electronic medical devices (e.g., cochlear implants, vagus nerve stimulator)
4. History of chronic pain previous to the amputation.
5. Head injury resulting in loss of consciousness for at least 30 min or pos-traumatic amnesia for greater than 24 hours, as self-reported
6. Unstable medical conditions (e.g. uncontrolled diabetes, uncompensated cardiac issues, heart failure or chronic obstructive pulmonary disease).
7. Uncontrolled Epilepsy or prior seizures within the last 1 year.
8. Suffering from severe depression (as defined by a score of >30 in the Beck Depression Inventory).*
9. History of unexplained fainting spells or loss of consciousness as self-reported during the last 2 years.
10. History of neurosurgery, as self-reported.
11. Mirror Therapy in the previous 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2015-07; Primary Completion 2020-03-27 (Actual); Study Completion 2026-12-21 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Felipe Fregni, MD, PhD, MPH, Principal Investigator — Spaulding Rehabilitation Hospital
Locations (2):
- Spaulding Rehabilitation Network Research Institute, Charlestown, Massachusetts, United States
- IMREA HCFMUSP - Rede Lucy Montoro, São Paulo, Brazil

REFERENCES:
- [Background] Flor H. Phantom-limb pain: characteristics, causes, and treatment. Lancet Neurol. 2002 Jul;1(3):182-9. doi: 10.1016/s1474-4422(02)00074-1. PMID 12849487
- [Background] Nikolajsen L, Staehelin Jensen T. Phantom limb pain. Curr Rev Pain. 2000;4(2):166-70. doi: 10.1007/s11916-000-0052-0. PMID 10998730
- [Background] Manchikanti L, Singh V. Managing phantom pain. Pain Physician. 2004 Jul;7(3):365-75. PMID 16858476
- [Background] Birbaumer N, Lutzenberger W, Montoya P, Larbig W, Unertl K, Topfner S, Grodd W, Taub E, Flor H. Effects of regional anesthesia on phantom limb pain are mirrored in changes in cortical reorganization. J Neurosci. 1997 Jul 15;17(14):5503-8. doi: 10.1523/JNEUROSCI.17-14-05503.1997. PMID 9204932
- [Background] Borsook D, Becerra L, Fishman S, Edwards A, Jennings CL, Stojanovic M, Papinicolas L, Ramachandran VS, Gonzalez RG, Breiter H. Acute plasticity in the human somatosensory cortex following amputation. Neuroreport. 1998 Apr 20;9(6):1013-7. doi: 10.1097/00001756-199804200-00011. PMID 9601659
- [Background] Flor H, Elbert T, Knecht S, Wienbruch C, Pantev C, Birbaumer N, Larbig W, Taub E. Phantom-limb pain as a perceptual correlate of cortical reorganization following arm amputation. Nature. 1995 Jun 8;375(6531):482-4. doi: 10.1038/375482a0. PMID 7777055
- [Background] Grusser SM, Winter C, Muhlnickel W, Denke C, Karl A, Villringer K, Flor H. The relationship of perceptual phenomena and cortical reorganization in upper extremity amputees. Neuroscience. 2001;102(2):263-72. doi: 10.1016/s0306-4522(00)00491-7. PMID 11166112
- [Background] Montoya P, Ritter K, Huse E, Larbig W, Braun C, Topfner S, Lutzenberger W, Grodd W, Flor H, Birbaumer N. The cortical somatotopic map and phantom phenomena in subjects with congenital limb atrophy and traumatic amputees with phantom limb pain. Eur J Neurosci. 1998 Mar;10(3):1095-102. doi: 10.1046/j.1460-9568.1998.00122.x. PMID 9753177
- [Background] Ramachandran VS, Rogers-Ramachandran D, Stewart M. Perceptual correlates of massive cortical reorganization. Science. 1992 Nov 13;258(5085):1159-60. doi: 10.1126/science.1439826. No abstract available.
- [Background] Davis KD, Kwan CL, Crawley AP, Mikulis DJ. Event-related fMRI of pain: entering a new era in imaging pain. Neuroreport. 1998 Sep 14;9(13):3019-23. doi: 10.1097/00001756-199809140-00018. PMID 9804308
- [Background] Foell J, Bekrater-Bodmann R, Diers M, Flor H. Mirror therapy for phantom limb pain: brain changes and the role of body representation. Eur J Pain. 2014 May;18(5):729-39. doi: 10.1002/j.1532-2149.2013.00433.x. Epub 2013 Dec 10. PMID 24327313
- [Background] Lotze M, Flor H, Grodd W, Larbig W, Birbaumer N. Phantom movements and pain. An fMRI study in upper limb amputees. Brain. 2001 Nov;124(Pt 11):2268-77. doi: 10.1093/brain/124.11.2268. PMID 11673327
- [Background] Gandiga PC, Hummel FC, Cohen LG. Transcranial DC stimulation (tDCS): a tool for double-blind sham-controlled clinical studies in brain stimulation. Clin Neurophysiol. 2006 Apr;117(4):845-50. doi: 10.1016/j.clinph.2005.12.003. Epub 2006 Jan 19. PMID 16427357
- [Background] Bolognini N, Olgiati E, Maravita A, Ferraro F, Fregni F. Motor and parietal cortex stimulation for phantom limb pain and sensations. Pain. 2013 Aug;154(8):1274-80. doi: 10.1016/j.pain.2013.03.040. Epub 2013 Apr 19. PMID 23707312
- [Background] Bolognini N, Spandri V, Olgiati E, Fregni F, Ferraro F, Maravita A. Long-term analgesic effects of transcranial direct current stimulation of the motor cortex on phantom limb and stump pain: a case report. J Pain Symptom Manage. 2013 Oct;46(4):e1-4. doi: 10.1016/j.jpainsymman.2013.06.014. Epub 2013 Aug 7. No abstract available. PMID 23932177
- [Background] Facchini S, Romani M, Tinazzi M, Aglioti SM. Time-related changes of excitability of the human motor system contingent upon immobilisation of the ring and little fingers. Clin Neurophysiol. 2002 Mar;113(3):367-75. doi: 10.1016/s1388-2457(02)00009-3. PMID 11897537
- [Background] Rioult-Pedotti MS, Friedman D, Hess G, Donoghue JP. Strengthening of horizontal cortical connections following skill learning. Nat Neurosci. 1998 Jul;1(3):230-4. doi: 10.1038/678. PMID 10195148
- [Background] Boggio PS, Castro LO, Savagim EA, Braite R, Cruz VC, Rocha RR, Rigonatti SP, Silva MT, Fregni F. Enhancement of non-dominant hand motor function by anodal transcranial direct current stimulation. Neurosci Lett. 2006 Aug 14;404(1-2):232-6. doi: 10.1016/j.neulet.2006.05.051. Epub 2006 Jun 30. PMID 16808997
- [Background] Fregni F, Boggio PS, Mansur CG, Wagner T, Ferreira MJ, Lima MC, Rigonatti SP, Marcolin MA, Freedman SD, Nitsche MA, Pascual-Leone A. Transcranial direct current stimulation of the unaffected hemisphere in stroke patients. Neuroreport. 2005 Sep 28;16(14):1551-5. doi: 10.1097/01.wnr.0000177010.44602.5e. PMID 16148743
- [Background] Hummel F, Cohen LG. Improvement of motor function with noninvasive cortical stimulation in a patient with chronic stroke. Neurorehabil Neural Repair. 2005 Mar;19(1):14-9. doi: 10.1177/1545968304272698. PMID 15673839
- [Background] Floel A, Cohen LG. Contribution of noninvasive cortical stimulation to the study of memory functions. Brain Res Rev. 2007 Feb;53(2):250-9. doi: 10.1016/j.brainresrev.2006.08.006. Epub 2006 Oct 4. PMID 17023050
- [Background] Monti A, Cogiamanian F, Marceglia S, Ferrucci R, Mameli F, Mrakic-Sposta S, Vergari M, Zago S, Priori A. Improved naming after transcranial direct current stimulation in aphasia. J Neurol Neurosurg Psychiatry. 2008 Apr;79(4):451-3. doi: 10.1136/jnnp.2007.135277. Epub 2007 Dec 20. PMID 18096677
- [Background] Iyer MB, Mattu U, Grafman J, Lomarev M, Sato S, Wassermann EM. Safety and cognitive effect of frontal DC brain polarization in healthy individuals. Neurology. 2005 Mar 8;64(5):872-5. doi: 10.1212/01.WNL.0000152986.07469.E9. PMID 15753425
- [Background] Fregni F, Boggio PS, Nitsche M, Bermpohl F, Antal A, Feredoes E, Marcolin MA, Rigonatti SP, Silva MT, Paulus W, Pascual-Leone A. Anodal transcranial direct current stimulation of prefrontal cortex enhances working memory. Exp Brain Res. 2005 Sep;166(1):23-30. doi: 10.1007/s00221-005-2334-6. Epub 2005 Jul 6. PMID 15999258
- [Background] MacIver K, Lloyd DM, Kelly S, Roberts N, Nurmikko T. Phantom limb pain, cortical reorganization and the therapeutic effect of mental imagery. Brain. 2008 Aug;131(Pt 8):2181-91. doi: 10.1093/brain/awn124. Epub 2008 Jun 20. PMID 18567624
- [Background] Rothgangel AS, Braun SM, Beurskens AJ, Seitz RJ, Wade DT. The clinical aspects of mirror therapy in rehabilitation: a systematic review of the literature. Int J Rehabil Res. 2011 Mar;34(1):1-13. doi: 10.1097/MRR.0b013e3283441e98. PMID 21326041
- [Background] Chan BL, Witt R, Charrow AP, Magee A, Howard R, Pasquina PF, Heilman KM, Tsao JW. Mirror therapy for phantom limb pain. N Engl J Med. 2007 Nov 22;357(21):2206-7. doi: 10.1056/NEJMc071927. No abstract available. PMID 18032777
- [Background] Darnall BD, Li H. Home-based self-delivered mirror therapy for phantom pain: a pilot study. J Rehabil Med. 2012 Mar;44(3):254-60. doi: 10.2340/16501977-0933. PMID 22378591
- [Background] MacLachlan M, McDonald D, Waloch J. Mirror treatment of lower limb phantom pain: a case study. Disabil Rehabil. 2004 Jul 22-Aug 5;26(14-15):901-4. doi: 10.1080/09638280410001708913. PMID 15497919
- [Background] Kim SY, Kim YY. Mirror therapy for phantom limb pain. Korean J Pain. 2012 Oct;25(4):272-4. doi: 10.3344/kjp.2012.25.4.272. Epub 2012 Oct 4. PMID 23091690
- [Background] Soler MD, Kumru H, Pelayo R, Vidal J, Tormos JM, Fregni F, Navarro X, Pascual-Leone A. Effectiveness of transcranial direct current stimulation and visual illusion on neuropathic pain in spinal cord injury. Brain. 2010 Sep;133(9):2565-77. doi: 10.1093/brain/awq184. Epub 2010 Aug 4. PMID 20685806
- [Background] Fregni F, Boggio PS, Lima MC, Ferreira MJ, Wagner T, Rigonatti SP, Castro AW, Souza DR, Riberto M, Freedman SD, Nitsche MA, Pascual-Leone A. A sham-controlled, phase II trial of transcranial direct current stimulation for the treatment of central pain in traumatic spinal cord injury. Pain. 2006 May;122(1-2):197-209. doi: 10.1016/j.pain.2006.02.023. Epub 2006 Mar 27. PMID 16564618
- [Background] Cheatle MD. Depression, chronic pain, and suicide by overdose: on the edge. Pain Med. 2011 Jun;12 Suppl 2(Suppl 2):S43-8. doi: 10.1111/j.1526-4637.2011.01131.x. PMID 21668756
- [Background] Brodie EE, Whyte A, Niven CA. Analgesia through the looking-glass? A randomized controlled trial investigating the effect of viewing a 'virtual' limb upon phantom limb pain, sensation and movement. Eur J Pain. 2007 May;11(4):428-36. doi: 10.1016/j.ejpain.2006.06.002. Epub 2006 Jul 20. PMID 16857400
- [Background] Moseley GL. Graded motor imagery for pathologic pain: a randomized controlled trial. Neurology. 2006 Dec 26;67(12):2129-34. doi: 10.1212/01.wnl.0000249112.56935.32. Epub 2006 Nov 2. PMID 17082465
- [Background] Kooijman CM, Dijkstra PU, Geertzen JHB, Elzinga A, van der Schans CP. Phantom pain and phantom sensations in upper limb amputees: an epidemiological study. Pain. 2000 Jul;87(1):33-41. doi: 10.1016/S0304-3959(00)00264-5. PMID 10863043
- [Background] Whyte AS, Niven CA. Psychological distress in amputees with phantom limb pain. J Pain Symptom Manage. 2001 Nov;22(5):938-46. doi: 10.1016/s0885-3924(01)00352-9. PMID 11728797
- [Background] Villamar MF, Wivatvongvana P, Patumanond J, Bikson M, Truong DQ, Datta A, Fregni F. Focal modulation of the primary motor cortex in fibromyalgia using 4x1-ring high-definition transcranial direct current stimulation (HD-tDCS): immediate and delayed analgesic effects of cathodal and anodal stimulation. J Pain. 2013 Apr;14(4):371-83. doi: 10.1016/j.jpain.2012.12.007. Epub 2013 Feb 14. PMID 23415877
- [Background] Portilla AS, Bravo GL, Miraval FK, Villamar MF, Schneider JC, Ryan CM, Fregni F. A feasibility study assessing cortical plasticity in chronic neuropathic pain following burn injury. J Burn Care Res. 2013 Jan-Feb;34(1):e48-52. doi: 10.1097/BCR.0b013e3182700675. PMID 23292595
- [Background] Beck AT, Epstein N, Brown G, Steer RA. An inventory for measuring clinical anxiety: psychometric properties. J Consult Clin Psychol. 1988 Dec;56(6):893-7. doi: 10.1037//0022-006x.56.6.893. No abstract available. PMID 3204199
- [Background] Pangman VC, Sloan J, Guse L. An examination of psychometric properties of the mini-mental state examination and the standardized mini-mental state examination: implications for clinical practice. Appl Nurs Res. 2000 Nov;13(4):209-13. doi: 10.1053/apnr.2000.9231. PMID 11078787
- [Background] Aldington D, Small C, Edwards D, Ralph J, Woods P, Jagdish S, Moore RA. A survey of post-amputation pains in serving military personnel. J R Army Med Corps. 2014 Mar;160(1):38-41. doi: 10.1136/jramc-2013-000069. Epub 2013 Jul 13. PMID 24109094
- [Background] Rahimi A, Mousavi B, Soroush M, Masumi M, Montazeri A. Pain and health-related quality of life in war veterans with bilateral lower limb amputations. Trauma Mon. 2012 Summer;17(2):282-6. doi: 10.5812/traumamon.5135. Epub 2012 Jul 31. PMID 24350107
- [Background] Sinha R, van den Heuvel WJ, Arokiasamy P, van Dijk JP. Influence of adjustments to amputation and artificial limb on quality of life in patients following lower limb amputation. Int J Rehabil Res. 2014 Mar;37(1):74-9. doi: 10.1097/MRR.0000000000000038. PMID 24157864
- [Background] Ware JE Jr, Gandek B, Kosinski M, Aaronson NK, Apolone G, Brazier J, Bullinger M, Kaasa S, Leplege A, Prieto L, Sullivan M, Thunedborg K. The equivalence of SF-36 summary health scores estimated using standard and country-specific algorithms in 10 countries: results from the IQOLA Project. International Quality of Life Assessment. J Clin Epidemiol. 1998 Nov;51(11):1167-70. doi: 10.1016/s0895-4356(98)00108-5. PMID 9817134
- [Background] Chan EA, Chung JW, Wong TK, Lien AS, Yang JY. Application of a virtual reality prototype for pain relief of pediatric burn in Taiwan. J Clin Nurs. 2007 Apr;16(4):786-93. doi: 10.1111/j.1365-2702.2006.01719.x. PMID 17402961
- [Background] Baudic S, Attal N, Mhalla A, Ciampi de Andrade D, Perrot S, Bouhassira D. Unilateral repetitive transcranial magnetic stimulation of the motor cortex does not affect cognition in patients with fibromyalgia. J Psychiatr Res. 2013 Jan;47(1):72-7. doi: 10.1016/j.jpsychires.2012.09.003. Epub 2012 Oct 15. PMID 23079535
- [Background] Souto G, Borges IC, Goes BT, de Mendonca ME, Goncalves RG, Garcia LB, Sa KN, Coutinho MR, Galvao-Castro B, Fregni F, Baptista AF. Effects of tDCS-induced motor cortex modulation on pain in HTLV-1: a blind randomized clinical trial. Clin J Pain. 2014 Sep;30(9):809-15. doi: 10.1097/AJP.0000000000000037. PMID 24300224
- [Background] Rossi S, Hallett M, Rossini PM, Pascual-Leone A; Safety of TMS Consensus Group. Safety, ethical considerations, and application guidelines for the use of transcranial magnetic stimulation in clinical practice and research. Clin Neurophysiol. 2009 Dec;120(12):2008-2039. doi: 10.1016/j.clinph.2009.08.016. Epub 2009 Oct 14. PMID 19833552
- [Background] Brunoni AR, Schestatsky P, Lotufo PA, Bensenor IM, Fregni F. Comparison of blinding effectiveness between sham tDCS and placebo sertraline in a 6-week major depression randomized clinical trial. Clin Neurophysiol. 2014 Feb;125(2):298-305. doi: 10.1016/j.clinph.2013.07.020. Epub 2013 Aug 30. PMID 23994192
- [Background] Klein MM, Treister R, Raij T, Pascual-Leone A, Park L, Nurmikko T, Lenz F, Lefaucheur JP, Lang M, Hallett M, Fox M, Cudkowicz M, Costello A, Carr DB, Ayache SS, Oaklander AL. Transcranial magnetic stimulation of the brain: guidelines for pain treatment research. Pain. 2015 Sep;156(9):1601-1614. doi: 10.1097/j.pain.0000000000000210. PMID 25919472
- [Background] Williams JA, Pascual-Leone A, Fregni F. Interhemispheric modulation induced by cortical stimulation and motor training. Phys Ther. 2010 Mar;90(3):398-410. doi: 10.2522/ptj.20090075. Epub 2010 Jan 28. PMID 20110339
- [Background] Rossini PM, Micera S, Benvenuto A, Carpaneto J, Cavallo G, Citi L, Cipriani C, Denaro L, Denaro V, Di Pino G, Ferreri F, Guglielmelli E, Hoffmann KP, Raspopovic S, Rigosa J, Rossini L, Tombini M, Dario P. Double nerve intraneural interface implant on a human amputee for robotic hand control. Clin Neurophysiol. 2010 May;121(5):777-83. doi: 10.1016/j.clinph.2010.01.001. Epub 2010 Jan 27. PMID 20110193
- [Background] Kujirai T, Sato M, Rothwell JC, Cohen LG. The effect of transcranial magnetic stimulation on median nerve somatosensory evoked potentials. Electroencephalogr Clin Neurophysiol. 1993 Aug;89(4):227-34. doi: 10.1016/0168-5597(93)90100-4. PMID 7688685
- [Background] Reuter M, Fischl B. Avoiding asymmetry-induced bias in longitudinal image processing. Neuroimage. 2011 Jul 1;57(1):19-21. doi: 10.1016/j.neuroimage.2011.02.076. Epub 2011 Mar 3. PMID 21376812
- [Background] Villiger M, Estevez N, Hepp-Reymond MC, Kiper D, Kollias SS, Eng K, Hotz-Boendermaker S. Enhanced activation of motor execution networks using action observation combined with imagination of lower limb movements. PLoS One. 2013 Aug 28;8(8):e72403. doi: 10.1371/journal.pone.0072403. eCollection 2013. PMID 24015241
- [Background] Iseki K, Hanakawa T, Shinozaki J, Nankaku M, Fukuyama H. Neural mechanisms involved in mental imagery and observation of gait. Neuroimage. 2008 Jul 1;41(3):1021-31. doi: 10.1016/j.neuroimage.2008.03.010. Epub 2008 Mar 20. PMID 18450480
- [Background] Bajwa S, Bermpohl F, Rigonatti SP, Pascual-Leone A, Boggio PS, Fregni F. Impaired interhemispheric interactions in patients with major depression. J Nerv Ment Dis. 2008 Sep;196(9):671-7. doi: 10.1097/NMD.0b013e318183f86f. PMID 18791428
- [Background] Schwenkreis P, Witscher K, Janssen F, Dertwinkel R, Zenz M, Malin JP, Tegenthoff M. Changes of cortical excitability in patients with upper limb amputation. Neurosci Lett. 2000 Oct 27;293(2):143-6. doi: 10.1016/s0304-3940(00)01517-2. PMID 11027854
- [Background] Moller HJ, Muller H, Borison RL, Schooler NR, Chouinard G. A path-analytical approach to differentiate between direct and indirect drug effects on negative symptoms in schizophrenic patients. A re-evaluation of the North American risperidone study. Eur Arch Psychiatry Clin Neurosci. 1995;245(1):45-9. doi: 10.1007/BF02191543. PMID 7540426
- [Background] Boynton GM, Engel SA, Glover GH, Heeger DJ. Linear systems analysis of functional magnetic resonance imaging in human V1. J Neurosci. 1996 Jul 1;16(13):4207-21. doi: 10.1523/JNEUROSCI.16-13-04207.1996. PMID 8753882
- [Background] Forman SD, Cohen JD, Fitzgerald M, Eddy WF, Mintun MA, Noll DC. Improved assessment of significant activation in functional magnetic resonance imaging (fMRI): use of a cluster-size threshold. Magn Reson Med. 1995 May;33(5):636-47. doi: 10.1002/mrm.1910330508. PMID 7596267
- [Background] Fregni F, Boggio PS, Nitsche MA, Marcolin MA, Rigonatti SP, Pascual-Leone A. Treatment of major depression with transcranial direct current stimulation. Bipolar Disord. 2006 Apr;8(2):203-4. doi: 10.1111/j.1399-5618.2006.00291.x. No abstract available. PMID 16542193
- [Background] Nitsche MA, Schauenburg A, Lang N, Liebetanz D, Exner C, Paulus W, Tergau F. Facilitation of implicit motor learning by weak transcranial direct current stimulation of the primary motor cortex in the human. J Cogn Neurosci. 2003 May 15;15(4):619-26. doi: 10.1162/089892903321662994. PMID 12803972
- [Background] Nitsche MA, Fricke K, Henschke U, Schlitterlau A, Liebetanz D, Lang N, Henning S, Tergau F, Paulus W. Pharmacological modulation of cortical excitability shifts induced by transcranial direct current stimulation in humans. J Physiol. 2003 Nov 15;553(Pt 1):293-301. doi: 10.1113/jphysiol.2003.049916. Epub 2003 Aug 29. PMID 12949224
- [Background] Nitsche MA, Liebetanz D, Antal A, Lang N, Tergau F, Paulus W. Modulation of cortical excitability by weak direct current stimulation--technical, safety and functional aspects. Suppl Clin Neurophysiol. 2003;56:255-76. doi: 10.1016/s1567-424x(09)70230-2. No abstract available. PMID 14677403
- [Background] Priori A. Brain polarization in humans: a reappraisal of an old tool for prolonged non-invasive modulation of brain excitability. Clin Neurophysiol. 2003 Apr;114(4):589-95. doi: 10.1016/s1388-2457(02)00437-6. PMID 12686266
- [Background] Nitsche MA, Liebetanz D, Lang N, Antal A, Tergau F, Paulus W. Safety criteria for transcranial direct current stimulation (tDCS) in humans. Clin Neurophysiol. 2003 Nov;114(11):2220-2; author reply 2222-3. doi: 10.1016/s1388-2457(03)00235-9. No abstract available. PMID 14580622
- [Background] Nitsche MA, Cohen LG, Wassermann EM, Priori A, Lang N, Antal A, Paulus W, Hummel F, Boggio PS, Fregni F, Pascual-Leone A. Transcranial direct current stimulation: State of the art 2008. Brain Stimul. 2008 Jul;1(3):206-23. doi: 10.1016/j.brs.2008.06.004. Epub 2008 Jul 1. PMID 20633386
- [Background] Nitsche MA, Jaussi W, Liebetanz D, Lang N, Tergau F, Paulus W. Consolidation of human motor cortical neuroplasticity by D-cycloserine. Neuropsychopharmacology. 2004 Aug;29(8):1573-8. doi: 10.1038/sj.npp.1300517. PMID 15199378
- [Background] Schley MT, Wilms P, Toepfner S, Schaller HP, Schmelz M, Konrad CJ, Birbaumer N. Painful and nonpainful phantom and stump sensations in acute traumatic amputees. J Trauma. 2008 Oct;65(4):858-64. doi: 10.1097/TA.0b013e31812eed9e. PMID 18849803
- [Background] Fregni F, Gimenes R, Valle AC, Ferreira MJ, Rocha RR, Natalle L, Bravo R, Rigonatti SP, Freedman SD, Nitsche MA, Pascual-Leone A, Boggio PS. A randomized, sham-controlled, proof of principle study of transcranial direct current stimulation for the treatment of pain in fibromyalgia. Arthritis Rheum. 2006 Dec;54(12):3988-98. doi: 10.1002/art.22195. PMID 17133529
- [Background] CREUTZFELDT OD, FROMM GH, KAPP H. Influence of transcortical d-c currents on cortical neuronal activity. Exp Neurol. 1962 Jun;5:436-52. doi: 10.1016/0014-4886(62)90056-0. No abstract available. PMID 13882165
- [Background] Wassermann EM. Risk and safety of repetitive transcranial magnetic stimulation: report and suggested guidelines from the International Workshop on the Safety of Repetitive Transcranial Magnetic Stimulation, June 5-7, 1996. Electroencephalogr Clin Neurophysiol. 1998 Jan;108(1):1-16. doi: 10.1016/s0168-5597(97)00096-8. PMID 9474057
- [Derived] Pinto CB, Saleh Velez FG, Bolognini N, Crandell D, Merabet LB, Fregni F. Optimizing Rehabilitation for Phantom Limb Pain Using Mirror Therapy and Transcranial Direct Current Stimulation: A Randomized, Double-Blind Clinical Trial Study Protocol. JMIR Res Protoc. 2016 Jul 6;5(3):e138. doi: 10.2196/resprot.5645. PMID 27383993

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Please note that from 132 subjects enrolled, 112 started (were randomized) as 20 subjects screened out after signing the consent form (time commitment=8; loss of interest=5; no more phantom limb pain=3; personal reasons=4).
Period: Overall Study
Arm/Group | Active tDCS and Active Mirror Therapy | Active tDCS and Sham Mirror Therapy | Sham tDCS and Active Mirror Therapy | Sham tDCS and Sham Mirrory Therapy
Started | 29 | 28 | 28 | 27
Completed | 28 | 24 | 26 | 25
Not Completed | 1 | 4 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active tDCS and Active Mirror Therapy | Active tDCS and Sham Mirror Therapy | Sham tDCS and Active Mirror Therapy | Sham tDCS and Sham Mirrory Therapy | Total
Number analyzed (Participants) | 29 | 28 | 28 | 27 | 112
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.24 (16.28) | 39.96 (15.96) | 46 (12.73) | 42.96 (12.28) | 44.34 (14.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 10 | 11 | 10 | 38
  Male | 22 | 18 | 17 | 17 | 74
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 0 | 0 | 2
  Asian | 0 | 1 | 1 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 7 | 6 | 6 | 6 | 25
  White | 14 | 15 | 15 | 15 | 59
  More than one race | 4 | 5 | 5 | 5 | 19
  Unknown or Not Reported | 3 | 0 | 1 | 0 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10 | 9 | 10 | 10 | 39
  Brazil | 19 | 19 | 18 | 17 | 73
Phantom Limb Pain [Mean (Standard Deviation); unit: units on a scale] — This scale measures the severity of phantom limb pain as indexed by a Visual Analog Scale (VAS). The VAS pain scale is a simple 10- point scale (0 = ''no pain'', 10 = ''pain as bad as you can imagine'').
  units on a scale | 6.12 (1.88) | 6.29 (1.67) | 6.09 (1.75) | 5.90 (1.57) | 6.08 (1.71)

OUTCOME MEASURES:

1. Primary Outcome: Changes in the Visual Analog Scale for Phantom Limb Pain
Description: The primary endpoint will be the severity of pain measured by changes in PLP from baseline to 4 weeks (value at 4 weeks minus value at baseline), as indexed by a Visual Analog Scale (VAS). The VAS pain scale is a simple 10- point scale (0 = ''no pain'', 10 = ''pain as bad as you can imagine''). Since we are using a difference, smaller values (negative) represent a better outcome.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active tDCS and Active Mirror Therapy | Active tDCS and Sham Mirror Therapy | Sham tDCS and Active Mirror Therapy | Sham tDCS and Sham Mirrory Therapy
Number analyzed (Participants) | 29 | 28 | 28 | 27
units on a scale | -2.84 (2.95) | -3.35 (3.24) | -1.78 (2.96) | -2.58 (2.78)

2. Secondary Outcome: Changes in the Visual Analog Scale for Stump Pain
Description: The endpoint will be the severity of pain measured by changes in Stump Pain from baseline to 4 weeks (value at 4 weeks minus value at baseline), as indexed by a Visual Analog Scale (VAS). The VAS Phantom Limb Stump Pain scale is a simple 10- point scale (0 = ''no Phantom Limb Stump Pain'', 10 = ''Phantom Limb Stump Pain as bad as you can imagine''). Since we are using a difference, smaller values (negative) represent a better outcome.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active tDCS and Active Mirror Therapy | Active tDCS and Sham Mirror Therapy | Sham tDCS and Active Mirror Therapy | Sham tDCS and Sham Mirrory Therapy
Number analyzed (Participants) | 29 | 28 | 28 | 27
units on a scale | -1.31 (2.99) | -1.9 (3.99) | -0.91 (2.94) | -0.96 (2.84)

3. Secondary Outcome: Changes in the Visual Analog Scale for Phantom Limb Sensation
Description: The endpoint will be the severity of pain measured by changes in Phantom Limb Sensation from baseline to 4 weeks (value at 4 weeks minus value at baseline), as indexed by a Visual Analog Scale (VAS). The VAS Phantom Limb Sensation scale is a simple 10- point scale (0 = ''no Phantom Limb Sensation'', 10 = ''Phantom Limb Sensation as much as you can imagine''). Since we are using a difference, smaller values (negative) represent a better outcome.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active tDCS and Active Mirror Therapy | Active tDCS and Sham Mirror Therapy | Sham tDCS and Active Mirror Therapy | Sham tDCS and Sham Mirrory Therapy
Number analyzed (Participants) | 29 | 28 | 28 | 27
units on a scale | -1.86 (2.55) | -2.55 (2.64) | -1.35 (2.64) | -2.83 (3.87)

ADVERSE EVENTS:
Time Frame: 3 months
Description: adverse effects were collected with a questionnaire for adverse effects
Arm/Group | Active tDCS and Active Mirror Therapy | Active tDCS and Sham Mirror Therapy | Sham tDCS and Active Mirror Therapy | Sham tDCS and Sham Mirrory Therapy
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/28 | 0/28 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/28 | 0/28 | 0/27
Other Adverse Events (participants affected / at risk) | 7/29 | 6/28 | 6/28 | 6/27
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active tDCS and Active Mirror Therapy (N=29) | Active tDCS and Sham Mirror Therapy (N=28) | Sham tDCS and Active Mirror Therapy (N=28) | Sham tDCS and Sham Mirrory Therapy (N=27)
Tingling sensation over stimulation area (Skin and subcutaneous tissue disorders) | 7 (35) | 6 (32) | 6 (29) | 6 (30)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-14): https://cdn.clinicaltrials.gov/large-docs/66/NCT02487966/Prot_SAP_000.pdf